CLINICAL TRIAL: NCT02198833
Title: Clinical Study to Assess the Efficacy of a Novel Micro-Patterned Foley Catheter to Reduce Catheter-Associated UrinaryTract Infection Among Spinal Cord Injury Patients
Brief Title: Efficacy of Micro-Patterned Foley Catheter to Reduce Catheter-Associated Urinary Tract Infection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study catheter manufacturing issues. Poor enrollment.
Sponsor: Baylor College of Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rabih Darouiche, Physician, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SC120028; H-32673 (Other: Baylor College of Medicine)
Record Dates: First submitted 2014-07-21; First posted 2014-07-24 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Urinary Tract Infection
Keywords: Urinary Tract Infection; Bacteriuria; Transurethral Foley Catheter; Suprapubic Foley Catheter; Spinal Cord injury
MeSH Terms: conditions — Urinary Tract Infections; Bacteriuria; Spinal Cord Injuries | interventions — Microscopy, Electron, Scanning

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Micro-Patterned Foley Catheter (Experimental): Procedures: Foley Catheter Insertion, Device Specific Adverse Event Assessment, Urine Cultures, Foley Catheter Tip Culture, Scanning Electron Microscopy
  Interventions: Biological: Urine Culture; Device: Foley Catheter Tip Culture; Device: Scanning Electron Microscopy; Procedure: Device Specific Adverse Event Assessment; Procedure: Foley Catheter Insertion
- Standard-of-Care Foley Catheter (Active Comparator): Procedures: Foley Catheter Insertion, Device Specific Adverse Event Assessment, Urine Cultures, Foley Catheter Tip Culture, Scanning Electron Microscopy
  Interventions: Biological: Urine Culture; Device: Foley Catheter Tip Culture; Device: Scanning Electron Microscopy; Procedure: Device Specific Adverse Event Assessment; Procedure: Foley Catheter Insertion

INTERVENTIONS:
Biological: Urine Culture — Obtain urine culture every third day
Device: Foley Catheter Tip Culture — Catheter Tip Roll Plate Culture
Device: Scanning Electron Microscopy — Houston Site Only
Procedure: Device Specific Adverse Event Assessment — Assessment will be made of catheter patency and/or trauma related to catheter placement
Procedure: Foley Catheter Insertion — Insert Foley catheter for 15 day duration

SUMMARY:
The purpose of this study is to determine if the study Foley catheter with its patterned external surface can delay the time to the onset of urinary tract infection in spinal cord injury patients who are dependent on a Foley catheter for drainage of their urinary bladder.

DETAILED DESCRIPTION:
Roughly half of the two million nosocomial infections that occur each year are associated with the use of a medical device. Approximately 30 million urinary catheters are inserted each year into the bladder of over five million patients, and each catheterized patient is at risk of developing catheter-associated symptomatic urinary tract infection. About 95% of urinary tract infections are associated with the use of a urinary catheter. Not only is catheter associated urinary tract infection the most common nosocomial infection in general, but it is also the most common infectious reason for admission to the hospital among the population of 275 thousand Americans with spinal cord injury, which expands by approximately 12 thousand persons each year. Hospital-acquired infections boost today's healthcare costs by billions of dollars and healthcare providers are increasingly responsible for shouldering these costs.

Catheter-associated symptomatic urinary tract infection is usually caused by organisms that originate from the patient's own colonic and perineal flora, or the hands of healthcare personnel during catheter insertion and manipulation of the collection system. Microbial species predominantly migrate into the bladder extraluminally via the mucoid film that forms between the catheter surface and the urethra. Current approaches for preventing catheter-related infections include antimicrobial modification of the catheter surface. Although these antimicrobial-based catheters aim to eradicate bacteria residing in the vicinity of the catheter surface, they can result in antibiotic resistance, which could have serious implications on patient care.

A novel urinary catheter, the Micro-Patterned Foley catheter has been developed that incorporates a micro-pattern texture on the surface; the texture is too small to see or feel, but has demonstrated an impressive effect in the laboratory inhibiting microbial attachment to the surface and microbial migration along the micro-patterned catheter segments. The objective of the study is to determine whether the novel Micro-Patterned catheter can delay the onset of catheter associated urinary tract infection in catheterized spinal cord injured patients. If successful, this catheter will help improve quality of patient care and reduce cost of care by reducing the need for antibiotic treatment. This finding could extend to other patient populations that require urinary catheterization.

ELIGIBILITY:
Inclusion Criteria

* Veteran
* Hospitalized in one of the two participating Spinal Cord Injury Units
* Require a size 14, 16, or 18 French catheter
* Sign and date the written informed consent document acknowledging his/her desire to participate in the study, or if unable to sign due to spinal cord injury give verbal consent in front of two impartial witnesses who sign and date the informed consent document in the presence of the participant
* Be able to understand and comply with written and verbal protocol requirements, instructions, and protocol-stated restrictions
* Require insertion or exchange of a Foley catheter for no longer than 15 days.

Exclusion Criteria

* Unable to provide informed consent
* Has a current symptomatic urinary tract infection
* Has persistent bacteriuria that cannot be cleared with antimicrobial agents to a nominal level of less than 1,000 Colony Forming Units/mL prior to study catheter insertion
* Has a known bloodstream infection or an infection that requires prolonged antibiotic therapy
* Has periurethral inflammation or infection
* Has a known urethral anatomical anomaly which makes catheterization difficult
* Has a known silicone allergy or sensitivity
* Cannot accommodate a size 14,16 or 18 French Foley catheter.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rabih O Darouiche, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - James A. Haley Veterans' Hospital, Tampa, Florida
  - Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Number of patients entered in the study is too small for analysis of data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Micro-Patterned Foley Catheter | Standard-of-Care Foley Catheter
Started | 1 (Unable to clear urine of bacteria for all but one patient therefore catheter not placed) | 1 (Unable to clear urine of bacteria for all but one patient therefore catheter not placed.)
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No analysis completed due to inability to place study catheter in all but two patients due to inability to clear urine of bacteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Micro-Patterned Foley Catheter | Standard-of-Care Foley Catheter | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
  <=18 years |  |  | 0
  Between 18 and 65 years |  |  | 0
  >=65 years |  |  | 0
Age, Continuous
Sex: Female, Male
  Female |  |  | 0
  Male |  |  | 0
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Delay Onset of Catheter Associated Symptomatic Urinary Tract Infection
Description: Patients will be assessed daily for the occurrence of signs and symptoms of urinary tract infection. A single, independent evaluator (PI/co-investigator) will determine whether the subject has a catheter associated urinary tract infection based on pre-defined criteria that involve symptom reports and lab values without knowledge of or access to the catheter type randomly assigned to the patient.
Time Frame: 15 Days
Population: No analysis completed due to inability to place study catheter due to persistent bacterial colonization.
Arm/Group | Micro-Patterned Foley Catheter | Standard-of-Care Foley Catheter
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time to Occurrence of Asymptomatic Bacteruria or Funguria
Description: Urine cultures will be obtained every third day to assess for the presence of microbial growth.
Time Frame: 15 days
Population: No analysis completed. Study catheter placed in only 2 patients due to inability to clear bacterial from urinary bladder during screening.
Arm/Group | Micro-Patterned Foley Catheter | Standard-of-Care Foley Catheter
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Assess the Microbial Coverage and Biofilm Formation on Catheter Surface
Description: Catheters will be cultured by Roll-plate method for microbial growth. Catheters removed at the Houston site will also be evaluated by scanning electron microscopy to determine microbial coverage and biofilm formation.
Time Frame: Day 15 or upon removal of Foley Catheter
Population: as for outcome 2
Arm/Group | Micro-Patterned Foley Catheter | Standard-of-Care Foley Catheter
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Device Specific Adverse Event Assessments
Description: Patient will be assessed daily for signs and symptoms of infection. Catheter placement and patency will be confirmed. Insertion site will be evaluated for signs of inflammation and or trauma.
Time Frame: 15 Days
Population: as for outcome 2
Arm/Group | Micro-Patterned Foley Catheter | Standard-of-Care Foley Catheter
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse events for a one month period.
Description: Definitions of adverse events planned for use in this study did not differ from those of clinicaltrials.gov.
Arm/Group | Micro-Patterned Foley Catheter | Standard-of-Care Foley Catheter
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Two major factors: 1) Production of the study catheter took much longer than expected. Only size 16 French Foley available; and 2) The inability to clear asymptomatic bacteriuria from patients' urinary bladder prior to study catheter placement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No